CLINICAL TRIAL: NCT04220398
Title: A Prospective, Multicenter, Three-arm, Randomized, Controlled Study Comparing the Efficacy of Neoadjuvant Hormonal Therapy Combined With Systemic Chemotherapy (NCHT), Neoadjuvant Hormonal Therapy (NHT) and Radical Prostatectomy Only in Locally Advanced Prostate Cancer
Brief Title: Neoadjuvant Chemo-hormonal Therapy Combined With Radical Prostatectomy for Locally Advanced Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCANT-20
Record Dates: First submitted 2020-01-02; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer; Chemotherapy Effect; Hormone Sensitive Prostate Cancer; Locally Advanced Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized 2:2:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NCHT Group (Experimental): Neoadjuvant chemotherapy combined with hormone therapy, Radical Prostatectomy (RP)+ extended lymph node dissection
  Interventions: Drug: Neoadjuvant chemotherapy combined with hormone therapy; Procedure: Radical Prostatectomy (RP)+ extended lymph node dissection
- NHT Group (Active Comparator): Neoadjuvant hormonal therapy, radical Prostatectomy (RP)+ extended lymph node dissection.
  Interventions: Drug: Neoadjuvant hormone therapy; Procedure: Radical Prostatectomy (RP)+ extended lymph node dissection
- RP Group (Other): Radical Prostatectomy (RP)+ extended lymph node dissection alone.
  Interventions: Procedure: Radical Prostatectomy (RP)+ extended lymph node dissection

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy combined with hormone therapy — Docetaxel 75mg/m2 IV (every 3 weeks) +Prednisone 5mg BID orally + HT (Bicalutamide Tablets, 50mg QD orally; Goserelin, 3.6mg, subcutaneous injection, q28d), 4-6 cycles
  Other Names: NCHT
  Arms: NCHT Group
Drug: Neoadjuvant hormone therapy — HT (Bicalutamide Tablets, 50mg QD orally; Goserelin, 3.6mg, subcutaneous injection, q28d), 3-6 cycles
  Other Names: NHT
  Arms: NHT Group
Procedure: Radical Prostatectomy (RP)+ extended lymph node dissection — Radical Prostatectomy (RP)+ extended lymph node dissection: Within three months after neoadjuvant treatment.
  Treatment after prostatectomy: There will not have any drug treatment after surgery until disease progression.
  Pelvic lymph node dissection is required to reach the level of bilateral iliac artery. If the postoperative pathology indicated positive incisional margin or pelvic lymph node metastasis, pelvic adjuvant radiotherapy should be performed within 3 months after surgery.
  Other Names: RP+ePLND

SUMMARY:
To evaluate of the value of radical prostatectomy and extended pelvic lymph node dissection in locally advanced prostate cancer after neoadjuvant hormonal therapy with or without docetaxel chemotherapy.

DETAILED DESCRIPTION:
Using larger sample prospective randomized controlled study design, and comparing neoadjuvant HT combined with docetaxel chemotherapy to neoadjuvant HT followed by RP and extended lymph node dissection to determine whether neoadjuvant HT combined with docetaxel chemotherapy can more effectively improve biochemical progression-free survival of locally advanced prostate cancer patients.

Further analysis was performed to determine whether the treatment regimen helped to prolong the radiologic progression-free survival (rPFS) or OS in these patients.

The pathological changes of tumor before and after neoadjuvant treatment were also analyzed. To search for the important risk factors influencing the long-term prognosis of these patients, the safety characteristics of patients in different treatment groups were analyzed. Therefore, it can provide the basis for the formulation of the optimal treatment plan for locally advanced prostate cancer, prolong the survival time of patients and improve the quality of life.

Study design: Prospective，Multicenter, Open-label, Parallel group, Randomized (2:2:1) Controlled , Clinical Trial

Study group: Newly diagnosed, untreated cT3a-cT4 or any cT, cN1 in locally advanced hormone-sensitive prostate cancer.

Study group number: 475 cases, Randomized 2:2:1

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ Aged <75 years, male;
2. Histology or cytology diagnosis: Prostate adenocarcinoma;
3. ECOG performance Status ≤1; Expected lifetime ≥10 years;
4. Without clinical or radiographic metastases in 6 months (Bone scan, MRI or pelvic enhanced CT scan, PET-CT) before randomized;
5. The patients of locally advanced prostate cancer need to satisfy at least one of the following requirements: clinical stageT3a-T4, N0, M0; any T, N1, M0;
6. Without Androgen Blockade Treatment in 4 weeks before randomized;
7. Without radiographic treatment towards primary tumour;
8. Without opioids (including codeine and dextropropoxyphene) relieving relevant pain of cancer;
9. Without azole drugs (such as fluconazole, itraconazole);
10. Important laboratory indicators are as follows:

    1. Haemoglobin ≥90g/L
    2. ANC ≥ 1500/μL
    3. PLT≥100*10^9/L
    4. K+≥3.5mmol/L
    5. AST or ALT ≤1.5 times upper limit of normal (ULN), TBIL should be ≤ULN (except patients with certified Gilbert syndrome) and ALP≤5ULN
    6. ALB≥30g / L
    7. calculated Ccr>60 ml/min, serum creatinine ≤ ULN
11. Without swallowing disease, able to swallow the whole piece of drugs;
12. Without other tumour chemotherapy history, without chemotherapy and endocrine therapy contraindications;
13. If patient's spouse is at her childbearing age, the patient needs to agree that effective contraception should be taken during the treatment and 4 months after the operation.
14. Subjects volunteer to participate, the subject must sign an informed consent form (ICF), indicating the understanding of the purpose and the required procedures of the study, and willing to participate in the study. Subjects must be willing to comply with the prohibitions and restrictions set forth in the program.

Exclusion Criteria:

1. The pathology result of prostate is neuroendocrine prostate cancer, including small cell carcinoma;
2. Previous cytotoxic chemotherapy or biological therapy for prostate cancer;
3. Contraindications to prednisone, such as active infections or other disorders;
4. Patients with chronic disease needed to be given dose of prednisone (each time 5mg, bid a day) exceed the dose in the study;
5. High blood pressure with poor control of drugs (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥95mmHg);
6. Active or symptomatic viral hepatitis or other chronic liver disease, known infected with human immunodeficiency virus (HIV);
7. A disease history of pituitary or adrenal dysfunction;
8. Patients with active autoimmune disease who need hormone therapy;
9. Heart disease with clinical significance, including: myocardial infarction or arterial thrombosis occurred in the past 6 months; severe or unstable angina; New York Heart Association grade III or IV heart disease (Appendix 4); atrial fibrillation or other arrhythmias that require treatment;
10. Subjects who participated in other clinical studies within a month before the first use of chemotherapy; (the elution time is at least 5 times the half-life time of the study drug if the half-life time is too long.)
11. Patients with a history of hypersensitivity to Taxanes or docetaxel
12. Patients who are concomitantly receiving strong CYP3A4 inhibitors
13. Other circumstances considered inappropriate by investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
bPFS (Biochemical progression-free survival) | about 2 years
  Biochemical recurrence-free survival (bPFS): defined as the time from randomization to biochemical recurrence. The definition of biochemical recurrence is as follows: in the case of normal testosterone levels, the PSA was >0.2 ng/ml twice for more than 4 consecutive weeks.

SECONDARY OUTCOMES:
The 1-year biochemical progression-free survival (bPFS) rate | 1 year
  The ratio of patients whose consecutive postoperative PSA <0.2ng/ml within 1-year.
Overall survival (OS) | 5-10 years
  The time from randomization to death due to all causes.
Radiographic progression-free survival (rPFS) | 3-5 years
  The time from randomization to first confirmed imaging progression or death (whichever first is counted). Imaging progression was defined as one of the following: a. Progression of soft tissue lesions as defined in the revised RECIST 1.1 (Appendix 8) found by CT or MRI. b. Confirmation of bone metastasis lesions by ECT or PET-CT examination.
TTPP | 1-3 years
  The time from randomization to the time when PSA increased by 25%.
ECOG score progression-free survival | 3-5 years
  The time from treatment to the time of ECOG score progression.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Qi D, Wu C, Liu F, Gu K, Shi Z, Lin X, Tao S, Xu W, Brendler CB, Zheng Y, Xu J. Trends of prostate cancer incidence and mortality in Shanghai, China from 1973 to 2009. Prostate. 2015 Oct;75(14):1662-8. doi: 10.1002/pros.23046. Epub 2015 Jul 17. PMID 26184773
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Peyromaure M, Debre B, Mao K, Zhang G, Wang Y, Sun Z, Xu D, Jiang J, Sun Y. Management of prostate cancer in China: a multicenter report of 6 institutions. J Urol. 2005 Nov;174(5):1794-7. doi: 10.1097/01.ju.0000176817.46279.93. PMID 16217289
- [Background] Spahn M, Joniau S, Gontero P, Fieuws S, Marchioro G, Tombal B, Kneitz B, Hsu CY, Van Der Eeckt K, Bader P, Frohneberg D, Tizzani A, Van Poppel H. Outcome predictors of radical prostatectomy in patients with prostate-specific antigen greater than 20 ng/ml: a European multi-institutional study of 712 patients. Eur Urol. 2010 Jul;58(1):1-7; discussion 10-1. doi: 10.1016/j.eururo.2010.03.001. Epub 2010 Mar 17. PMID 20299147
- [Background] Eggener SE, Scardino PT, Walsh PC, Han M, Partin AW, Trock BJ, Feng Z, Wood DP, Eastham JA, Yossepowitch O, Rabah DM, Kattan MW, Yu C, Klein EA, Stephenson AJ. Predicting 15-year prostate cancer specific mortality after radical prostatectomy. J Urol. 2011 Mar;185(3):869-75. doi: 10.1016/j.juro.2010.10.057. Epub 2011 Jan 15. PMID 21239008
- [Background] Sfoungaristos S, Kourmpetis V, Fokaefs E, Perimenis P. Neoadjuvant Chemotherapy prior to Radical Prostatectomy for Patients with High-Risk Prostate Cancer: A Systematic Review. Chemother Res Pract. 2013;2013:386809. doi: 10.1155/2013/386809. Epub 2013 Feb 21. PMID 23509625
- [Background] Ward JF, Slezak JM, Blute ML, Bergstralh EJ, Zincke H. Radical prostatectomy for clinically advanced (cT3) prostate cancer since the advent of prostate-specific antigen testing: 15-year outcome. BJU Int. 2005 Apr;95(6):751-6. doi: 10.1111/j.1464-410X.2005.05394.x. PMID 15794776
- [Background] Shelley MD, Kumar S, Coles B, Wilt T, Staffurth J, Mason MD. Adjuvant hormone therapy for localised and locally advanced prostate carcinoma: a systematic review and meta-analysis of randomised trials. Cancer Treat Rev. 2009 Nov;35(7):540-6. doi: 10.1016/j.ctrv.2009.05.001. Epub 2009 Jun 2. PMID 19493624
- [Background] Hu J, Xu H, Zhu W, Wu F, Wang J, Ding Q, Jiang H. Neo-adjuvant hormone therapy for non-metastatic prostate cancer: a systematic review and meta-analysis of 5,194 patients. World J Surg Oncol. 2015 Feb 22;13:73. doi: 10.1186/s12957-015-0503-z. PMID 25884478
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Thalgott M, Horn T, Heck MM, Maurer T, Eiber M, Retz M, Autenrieth M, Herkommer K, Krause BJ, Gschwend JE, Treiber U, Kubler HR. Long-term results of a phase II study with neoadjuvant docetaxel chemotherapy and complete androgen blockade in locally advanced and high-risk prostate cancer. J Hematol Oncol. 2014 Mar 5;7:20. doi: 10.1186/1756-8722-7-20. PMID 24598155
- [Background] Prayer-Galetti T, Sacco E, Pagano F, Gardiman M, Cisternino A, Betto G, Sperandio P. Long-term follow-up of a neoadjuvant chemohormonal taxane-based phase II trial before radical prostatectomy in patients with non-metastatic high-risk prostate cancer. BJU Int. 2007 Aug;100(2):274-80. doi: 10.1111/j.1464-410X.2007.06760.x. Epub 2007 Mar 12. PMID 17355369
- [Background] Sella A, Zisman A, Kovel S, Yarom N, Leibovici D, Lindner A. Neoadjuvant chemohormonal therapy in poor-prognosis localized prostate cancer. Urology. 2008 Feb;71(2):323-7. doi: 10.1016/j.urology.2007.08.060. PMID 18308112

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT04220398/Prot_SAP_000.pdf